CLINICAL TRIAL: NCT00323440
Title: Inflammatory Proteins in Familial Mediterranean Fever During Attack and Remission
Status: Withdrawn | Type: Observational
Why Stopped: Collaboration could not be established
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-06-4126-AL-CTIL
Record Dates: First submitted 2006-05-07; First posted 2006-05-09 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Familial Mediterranean Fever
Keywords: Familial Mediterranean fever; Inflammation; Attacks; Remission; RNA; Cytokines; Inflammatory proteins; MEFV; mutations; Colchicine; Treatment; microarray RNA analysis
MeSH Terms: conditions — Familial Mediterranean Fever; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Group 1: FMF patients in remission
- Group 2: FMF patients during attack
- Group 3: FMF patients without colchicine in remission
- Group 4: FMF patients without colchicine in attack

SUMMARY:
Familial Mediterranean fever (FMF) is a genetic disease, caused by mutations in the FMF gene, entitled MEFV. The disease is characterized by painful attacks of inflammation in sites lined by serous membranes (e.g. abdominal pain caused by inflammation of the peritoneum, a serous membrane surrounding all internal organs within the abdomen). Continuous colchicine treatment prevents attacks in most patients. The pathogenesis of the disease, what leads to the attacks and how colchicine helps, are questions not yet resolved. Elucidating the role of the inflammatory proteins is an important step towards the understanding of these questions. To date only small numbers of cytokines and inflammatory proteins have been studied individually. We propose to study a large number of these proteins in the RNA and protein levels addressing the interaction between them and the effect of colchicine on their expression.

Blood samples will be drawn from consenting patients in remission, during attacks, under and without colchicine treatment. (20 patients in each category).Twenty healthy volunteers will donate control blood samples for the study. RNA will be produced from the neutrophils, and cytokines and various proteins' RNA expression will be determined. Major expressed proteins will be measured in the same samples and the results will be analyzed with regard to the activity of the disease, MEFV mutations and colchicine treatment status. The information obtained by the study may allow us to determine the sequence of events associated with FMF attack development, and perhaps take us one step further in the understanding of the pathogenesis of the disease.

DETAILED DESCRIPTION:
Familial Mediterranean fever (FMF) is a genetic disease, caused by mutations in the FMF gene, entitled MEFV. The disease is characterized by painful attacks of inflammation in sites lined by serous membranes (e.g. abdominal pain caused by inflammation of the peritoneum, a serous membrane surrounding all internal organs within the abdomen). Continuous colchicine treatment prevents attacks in most patients. The pathogenesis of the disease, what leads to the attacks and how colchicine helps, are questions not yet resolved. Elucidating the role of the inflammatory proteins is an important step towards the understanding of these questions. To date only small numbers of cytokines and inflammatory proteins have been studied individually. We propose to study a large number of these proteins in the RNA and protein levels addressing the interaction between them and the effect of colchicine on their expression.

Blood samples will be drawn from consenting patients in remission, during attacks, under and without colchicine treatment. (20 patients in each category).Twenty healthy volunteers will donate control blood samples for the study. RNA will be produced from the neutrophils, and cytokines and various proteins' RNA expression will be determined. Major expressed proteins will be measured in the same samples and the results will be analyzed with regard to the activity of the disease, MEFV mutations and colchicine treatment status. The information obtained by the study may allow us to determine the sequence of events associated with FMF attack development, and perhaps take us one step further in the understanding of the pathogenesis of the disease.

ELIGIBILITY:
Inclusion Criteria:

* FMF patients, agreeing with diagnostic criteria, in attack or remission, under or without colchicine treatment.
* Age 18 or older
* Male or female
* all ethnic groups arriving for treatment or routine follow up appointment
* Written Consent to participate and donate blood for protein, RNA and DNA analyses.

Exclusion Criteria:

* Younger than 18
* Patients that use anti inflammatory medications, other than colchicine
* Patients who in addition to FMF suffer from another acute infectious or inflammatory disease
* Patients who in addition to FMF suffer from another chronic infectious or inflammatory or autoimmune disease.
* Amyloidosis
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: FMF patients recruited at clinic on follow-up visits and FMF patients arriving at ER during attacks
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-08 (Estimated); Primary Completion 2010-08 (Estimated); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Avi Livneh, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel